CLINICAL TRIAL: NCT00056134
Title: Vaccination of HLA-A1 and/or -A2+ Stage III or IV Melanoma Patients With Tumor Peptide-Loaded Autologous Dendritic Cells With Prior Depletion of CD25-Positive Cells Using Denileukin Difitox (ONTAK)
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, PD Dr. med. univ. Beatrice Schuler-Thurner, Principal Investigator, University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000270762; ERLANGEN-ONTAK; EU-20246
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Dendritic cell vaccine plus denileukin difitox

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells mixed with tumor proteins may make the body build an immune response to kill tumor cells. Biological therapies such as denileukin diftitox may be able to deliver cancer-killing substances directly to melanoma cells. Combining vaccine therapy with biological therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining vaccine therapy with denileukin diftitox in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of vaccination with autologous dendritic cells pulsed with tumor and influenza antigen peptides with or without ex vivo CD40-ligand and denileukin diftitox, in terms of tumor-specific T-cell response, in patients with HLA-A1- and/or HLA-A2.1-positive stage III or IV melanoma.
* Determine the safety and tolerability of these vaccinations in these patients.
* Determine tumor response in patients treated with these vaccinations.

OUTLINE:

* Phase I (Administration of denileukin diftitox and vaccinations #1 to #4): Patients undergo leukapheresis for collection of peripheral blood mononuclear cells (PMBC). PBMC are processed for the generation of dendritic cells (DC) to be used for vaccinations. DC are pulsed with HLA-A1- and HLA-A2.1-restricted peptides derived from melanoma-associated tumor antigens. DC are pulsed with or without ex vivo treatment with CD40-ligand. Patients receive denileukin diftitox IV for 3 consecutive days before the first vaccination. Patients receive 4 pulsed DC vaccinations subcutaneously (SC) on days 1, 14, 42, and 70 in the absence of disease progression or unacceptable toxicity.

Patients who show a tumor response (at least stable disease) may receive vaccination #5 and further booster vaccinations.

* Phase II: DC are generated and pulsed as in phase I. Patients receive up to 6 additional booster pulsed DC vaccinations SC on days 126, 184, 268, 356, 520, and 692 in the absence of disease progession or unacceptable toxicity.

Patients are followed for 10 years.

PROJECTED ACCRUAL: A total of 8-30 patients will be accrued for this study within 6-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locoregional or metastatic cutaneous malignant melanoma

  * Stage III or IV disease

    * Stage III: pT4b, N0, M0 (satellite metastases) or any pT, N1 or pT, N1 or N2a-c, M0 (lymph node metastases or in transit intralymphatic metastases)
    * Stage IV: any pT, N1-2, M1a-b
    * Surgically incurable
    * Incurable with standard treatment (i.e., localized chemotherapy/limb perfusion for stage III, systemic chemotherapy for stage IV)
* Unidimensionally or bidimensionally measurable disease by physical examination (e.g., cutaneous metastases) and/or non-invasive radiologic procedures NOTE: Stage III lesions may be measurable lymph nodes after incomplete resection and/or inoperable in transit metastases
* HLA-A1 and/or HLA-A2 expression by serologic HLA typing

  * HLA-A2.01 subtype must be confirmed by polymerase chain reaction on genomic DNA obtained from peripheral blood mononuclear cells
* No active CNS metastases

  * Previously treated CNS metastases (e.g., excision of a single metastasis) allowed if no active disease present by CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 6 months

Hematopoietic

* WBC greater than 2,500/mm^3
* Neutrophil count greater than 1,000/mm^3
* Lymphocyte count greater than 700/mm^3
* Platelet count greater than 75,000/mm^3
* Hemoglobin greater than 9 g/dL
* No bleeding disorders

Hepatic

* Bilirubin less than 2.0 mg/dL
* No hepatitis B or C

Renal

* Creatinine less than 2.5 mg/dL

Cardiovascular

* No clinically significant heart disease

Pulmonary

* No clinically significant respiratory disease

Immunologic

* No active systemic infection
* No immunodeficiency disease

  * No evidence of HIV-1, HIV-2, or human T-cell lymphocytic virus-1
* No active autoimmune disease including, but not limited to:

  * Lupus erythematosus
  * Autoimmune thyroiditis or uveitis
  * Multiple sclerosis
  * Inflammatory bowel disease NOTE: Vitiligo allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No organic brain syndrome or significant psychiatric abnormality that would preclude study participation and follow-up
* No contraindication to leukapheresis
* No other active malignant neoplasms

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior systemic immunotherapy
* No concurrent immunotherapy during and for 2 weeks after last vaccination

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior systemic chemotherapy (6 weeks for nitrosoureas [e.g., fotemustine])
* No concurrent chemotherapy during and for 2 weeks after last vaccination

Endocrine therapy

* No concurrent corticosteroids during and for 2 weeks after last vaccination

Radiotherapy

* No prior radiotherapy to the spleen
* Concurrent palliative radiotherapy allowed for selected metastases (e.g., pain or local complications such as compression)

Surgery

* See Disease Characteristics
* Recovered from prior surgery
* No prior splenectomy
* No prior organ allografts
* Concurrent surgery of selected metastases (e.g., pain or local complications such as compression) allowed

Other

* No other concurrent investigational drugs during and for 2 weeks after last vaccination
* No concurrent paramedical substance during and for 2 weeks after last vaccination
* No concurrent participation or intent to participate in another clinical trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-10; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by clinical and laboratory evaluation at every visit
Overall survival as assessed by clinical staging (CT scan and positron emission tomography [PET]) every 3 months

SECONDARY OUTCOMES:
Depletion of regulatory T-cells as assessed by tetramer stainings at every visit
Induction of antigen-specific immune responses as assessed by elispot and tetramer staining at every visit
Time to progression as assessed by clinical staging (CT scan and PET) every 3 months
Objective response rate as assessed by clinical staging (CT scan and PET) every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Schuler, Study Chair — Dermatologische Klinik MIT Poliklinik-Universitaetsklinikum Erlangen
Locations (1):
- Dermatologische Klinik mit Poliklinik - Universitaetsklinikum Erlangen, Erlangen, Germany

REFERENCES:
- [Derived] Baur AS, Lutz MB, Schierer S, Beltrame L, Theiner G, Zinser E, Ostalecki C, Heidkamp G, Haendle I, Erdmann M, Wiesinger M, Leisgang W, Gross S, Pommer AJ, Kampgen E, Dudziak D, Steinkasserer A, Cavalieri D, Schuler-Thurner B, Schuler G. Denileukin diftitox (ONTAK) induces a tolerogenic phenotype in dendritic cells and stimulates survival of resting Treg. Blood. 2013 Sep 26;122(13):2185-94. doi: 10.1182/blood-2012-09-456988. Epub 2013 Aug 19. PMID 23958949
- Available data/document: Publication — https://www.ncbi.nlm.nih.gov/pubmed/23958949 — Denileukin diftitox (ONTAK) induces a tolerogenic phenotype in dendritic cells and stimulates survival of resting Treg. Baur AS1, Lutz MB, Schierer S, Beltrame L, Theiner G, Zinser E, Ostalecki C, Heidkamp G, Haendle I, Erdmann M, Wiesinger M, Leisgang W, Gross S, Pommer AJ, Kämpgen E, Dudziak D, Steinkasserer A, Cavalieri D, Schuler-Thurner B, Schuler G.
- Available data/document: Clinical Study Report: DOI:10.1182/blood-2012-09-4569 — https://www.ncbi.nlm.nih.gov/pubmed/23958949 — Denileukin diftitox (ONTAK) induces... Baur AS et al